CLINICAL TRIAL: NCT06706960
Title: The Jugular Vein Ultrasonography for Hydration Assessment in Healthy Participants - The THAP Study
Brief Title: The Jugular Vein Ultrasonography for Hydration Assessment in Healthy Participants
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-01640; kt24Potasso
Record Dates: First submitted 2024-11-22; First posted 2024-11-27 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-12

CONDITIONS: Water Balance Disorders; Dehydration; Hypervolemia
Keywords: jugular vein pressure; internal jugular vein; non-invasive hydration status assessment; Hydration
MeSH Terms: conditions — Dehydration; Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: measurement of IJV-height — Protocol 1: IJV tapering portion is portrayed in a transverse view. With a skin marker, the IJV height is marked and measured as soon as IJV is smaller than CCA throughout the whole respiratory cycle.
  Protocol 2: IJV tapering portion is portrayed in a transverse view. With a skin marker, the IJV height is marked and measured as soon as IJV is completely collapsed throughout the whole respiratory cycle.
  Protocol 3: IJV tapering portion is portrayed in a longitudinal view. With a skin marker, the IJV height at the end of expiration is marked and measured at the following two positions:
  1. Measurement 1: at the very end of the tapering portion (collapsing point / top of pulsation).
  2. Measurement 2: at the beginning of the tapering portion (taper point).

SUMMARY:
The aim of this cross-sectional, descriptive analysis is to compare 3 different ultrasound-based protocols to measure the internal jugular vein pressure (uJVP) in healthy individuals.

DETAILED DESCRIPTION:
Proper hydration is crucial for health, and imbalances-like dehydration or fluid overload-can cause serious health problems including increased morbidity, hospitalization rate, and even mortality. Currently, assessing hydration is challenging, and there is no standardized method in clinical use.

Ultrasound (US) of the internal jugular vein (IJV) and ultrasound-guided estimation of jugular venous pressure (uJVP) is a promising, non-invasive method to assess the hydration status. Several measure methods have been described, however, there is no univocal protocol for US IJV-assessment.

In this study, three existing protocols including 4 measurements are compared to measure uJVP, which reflects the body's fluid balance. The study aims to find out which method is most accurate, easy to perform, and consistent when done by the same or different medical professionals. They will also look at how long each method takes and how acceptable these tests are to participants.

The study is performed in healthy individuals and all 4 measurements are applied cross-sectional during one visit. The whole ultrasound assessment will have a duration of maximum 45 minutes.

For all protocols, uJVP will be calculated by measuring with a ruler the vertical distance between IJV-height and sternal angle (cm) and then adding 5cm to this value.

Protocol 1: IJV tapering portion is portrayed in a transverse view. The IJV height is marked and measured as soon as IJV is smaller than Common Carotid Artery (CCA) throughout the whole respiratory cycle.

Protocol 2: IJV tapering portion is portrayed in a transverse view. The IJV height is marked and measured as soon as IJV is completely collapsed throughout the whole respiratory cycle.

Protocol 3: IJV tapering portion is portrayed in a longitudinal view. The IJV height at the end of expiration is marked and measured at the following two positions:

1. Measurement 1: at the very end of the tapering portion (collapsing point / top of pulsation).
2. Measurement 2: at the beginning of the tapering portion (taper point).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18 years or older, 15 women and 15 men.

Exclusion Criteria:

1. Major cardiovascular event in the last 3 months
2. Pregnant or lactating women
3. Heart failure of any grade
4. Kidney failure
5. Thrombosis V. jugularis interna
6. Atrial Fibrillation
7. Valves impairment
8. Uncontrolled Diabetes mellitus
9. Uncontrolled Diabetes insipidus (AVP resistance or deficiency)
10. Respiratory Distress of any grade
11. Signs/Symptoms of volume loss (diarrhea, vomiting, bleeding) in the past 3 days
12. Medication: Angiotensin-converting enzyme inhibitors, Angiotensin receptor blockers, any diuretic therapy
13. Inability to follow procedures or insufficient knowledge of project language.
14. Inability to give consent
15. Abnormal vital signs: tachycardia > 90/min, systolic blood pressure < 90 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment will take place at university hospital of Basel through flyers and word of mouth addressed to healthy visitors and employees.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Variance analysis | The whole ultrasound assessment will have a duration of maximum 45 minutes
  Percentage of participants differing > 1 Standard Deviation (SD) from the expected value of Ultrasound-guided Jugular Venous Pressure (uJVP) measured in cm for each of the 3 protocols

SECONDARY OUTCOMES:
Interpersonal variance analysis | The whole ultrasound assessment will have a duration of maximum 45 minutes
  Interpersonal variance analysis of the results for uJVP (cm) for each of the 3 different protocols, as well as for collapsibility index (%) and Jugular Vein Diameter (JVD) ratio
Intrapersonal variance analysis | The whole ultrasound assessment will have a duration of maximum 45 minutes
  Intrapersonal variance analysis of the results for uJVP (cm) for each of the 3 different protocols, as well as for collapsibility index (%) and JVD ratio
Timepoint-dependent Intrapersonal variance analysis | The whole ultrasound assessment will have a duration of maximum 45 minutes
  Intrapersonal variance analysis according to timepoint of US-assessment (first 15 participants vs last 15 participants)
Duration of the US assessment | The whole ultrasound assessment will have a duration of maximum 45 minutes
  Duration of the US assessment (minutes): interpersonal and intrapersonal variance analysis, protocol 1 vs 2 vs 3
Descriptive analysis | The whole ultrasound assessment will have a duration of maximum 45 minutes
  Descriptive analysis of analogue Visual Analogue Scale (VAS) Score data about acceptance of the 3 different US assessment protocols

CONTACTS AND LOCATIONS:
Overall Officials: Laura Potasso, Dr. med. sc., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No